CLINICAL TRIAL: NCT01220843
Title: Randomized Placebo Controlled Double-blind Trial in CKD Patients Not on Dialysis to Evaluate the Effect of Sevelamer Carbonate in the Control of FGF-23 Serum Levels and Its Consequences in the Evolution of PTH, Calcitriol and Mineral Metabolism Parameters Levels
Brief Title: FGF23 Reduction : Efficacy of a New Phosphate Binder in CHronic Kidney Disease
Acronym: FRENCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI10-PR-CHOUKROUN-1; 2010-020872-49 (EudraCT Number)
Record Dates: First submitted 2010-10-12; First posted 2010-10-14 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Chronic Renal Failure
Keywords: chronic renal failure; FGF23; Sevelamer carbonate
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Sevelamer

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): DOuble blinded, same labels than the active drug same dosage (2 tablets 3 times per day) during the meal
  Interventions: Drug: Placebo
- Sevelamer carbonate (Experimental): DOuble blinded, dosage 2 tablets 3 times per day corresponding to 4.8/d to taken during meals
  Interventions: Drug: Sevelamer carbonate

INTERVENTIONS:
Drug: Placebo — dosage : 2 tablets 3 times per day corresponding taken during meals during 12 weeks
  Arms: Placebo
Drug: Sevelamer carbonate — dosage : 2 tablets 3 times per day corresponding taken during meals during 12 weeks ( each tablet :800mg sevelamer carbonate
  Other Names: Renvela 800
  Arms: Sevelamer carbonate

SUMMARY:
The purpose of this study is to evaluate in Chronic Kidney Disease (CKD) patients not on dialysis and who have an Fibroblast growth factor 23 (FGF23) serum levels elevated, the effect of non calcic phosphate binder: sevelamer carbonate. This treatment could lead to a diminution of FGF23 serum levels due to the diminution of intestinal absorption of dietary phosphate. In addition, the investigators will describe the impact of the FGF23 level monitoring on the main phosphocalcium metabolism markers as phosphatemia, intact parathyroid hormone (iPTH), serum calcitriol and phosphaturia.

DETAILED DESCRIPTION:
The total length of the study is 14 weeks divided in 2 parts the first part is the screening period she will stay 1 to 2 weeks and the second period with the treatment with permanent dosage during 12 weeks.

During the screening visit (Vo) inclusion and non inclusion criteria will be checked and the patient consent will be collected. Biological analysis will be performed.

If the patient still eligible after the reception of biological results, he will be randomized and will received, either sevelamer carbonate, either placebo. The study treatment will be begun at the randomisation visit (V1) the dosage will be 2 tablets 3 times per day (corresponding to 4.8g/d sevelamer carbonate for patient taken active medication).

Patient will be seen every 2 weeks after the first visit (+/-5days) during 6 weeks (visit2/day15, visit3/day30, visit4/day45) and 12 weeks after the randomisation visit (visit5/day90). This visits will include biological analysis, compliance evaluation, adverse events report, concomitant treatments reports.

After the consent signature, all the adverse events will be collected until the end of the study for the patient (Visit5 or end of the study visit). Serious adverse events will be collected until 30 days after the date of the end of the study.

The same dosage of the study treatment will be followed during all the study period except if the phosphatemia (evaluated during one analysis) is found above the normal range planned by the protocol. In this case, the dosage adaptations will be :

* If during a visit the phosphatemia is above or equal to 0.8 mmol/l and superior to 0.5 mmol/l, the study treatment dosage need to be reduce to 2 tablets 3 times per day to 1 tablet 3 times per day.
* If during the next blood punction, the phosphatemia still or equal to 0.8 mmol/l and superior to 0.5 mmol/l, the study treatment will be stopped and a "end of study" visit will be performed.
* If during one study visit, the phosphatemia is above or equal to 0.5 mmol/l,the study treatment will be stopped immediately and a end of study visit will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who gave their written consent
* Women or men over 18 years
* No concomitant treatment with phosphate binders
* CKD patients not on dialysis stage 3b or 4, as a GFR (glomerular filtration rate) between 15 and 45 ml/min/1.73m2, using simplified MDRD formula
* At the inclusion visit,patients with blood results as levels of C-terminal FGF-23 > 120 rU/ml and fasting phosphatemia > 1.0 mmol/l
* Able to comply with the study procedures during all the study period
* Willing to abstain from taking any following medication during all the study period :antiacid and phosphate binders with aluminium, magnesium, calcium or lanthanum;Treatment for hyperparathyroid : active vitamin D and calcimimetic ; native vitamin D
* Female subjects who are of childbearing potential must have a reliable contraceptive methods during all the study period (hormonal, barrier methods or intrauterine device)
* No Participation in any clinical trial using an investigational product or device during the 30 days preceding the first protocol visit
* Informed patient who agreed with the utilisation of his data for the study
* Able to read and understand french and study objectives
* Inscription to medical assurance

Exclusion Criteria:

* predisposition with or presence of intestinal or ileus obstruction or severe gastrointestinal motility disorder(like severe constipation)
* Antecedent of major gastrointestinal surgery
* Abusive consumption of alcohol and drug (exclude tabacco) according the investigator
* Arrythmia treated by antiarrythmic agent or epilepsia treated by anticonvulsant
* Antecedent of kidney transplantation
* Antecedent of parathyroidectomy
* At the inclusion visit,patients with blood results as fasting phosphatemia > 1.78 mmol/l or serum 25(OH)D3< 20 ng/ml (<50 nmol/)
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2010-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Measurement of the serum levels of C terminal segment of fibroblast growth factor 23 (FGF23) and evaluation of sevelamer carbonate effect on this levels in comparison with placebo | 12 weeks after the beginning of treatment
  Indeed the sevelamer carbonate could lead to a diminution of FGF23 serum levels due to the diminution of intestinal absorption of dietary phosphate.

SECONDARY OUTCOMES:
Evaluation of sevelamer carbonate effect on the serum levels of iPTH | 12 weeks after the beginning of treatment
Evaluation of sevelamer carbonate effect on the serum levels of calcitriol (1 25(OH)2D3) | 12 weeks after the beginning of treatment
Evaluation of sevelamer carbonate effect on the serum levels of others mineral metabolism parameters (phosphore, calcium, intact FGF-23 , 25(OH)D3, bone specific alkaline phosphatases, osteocalcin, collagen crosslink, C reactive protein) | 12 weeks after the beginning of treatment
Evaluation of sevelamer carbonate effect on the urinary levels of phosphate | 12 weeks after the beginning of treatment
Evaluation of sevelamer carbonate effect on the urinary levels of calcium | 12 weeks after the beginning of treatment
Evaluation of sevelamer carbonate effect on the urinary levels of creatinine | 12 weeks after the beginning of treatment
Evaluation of sevelamer carbonate effect on the urinary levels of urea | 12 weeks after the beginning of treatment
Evaluation of sevelamer carbonate effect on the serum and urinary levels of specific biomarkers (serum : fetuin A, para-cresyl sulfate, osteopontin) | 12 weeks after the beginning of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Choukroun, Ph D, M D, Principal Investigator — Centre Hospitalier Universitaire, Amiens
Locations (15):
- France (15):
  - CHU Amiens service de nephrologie, Amiens
  - CHU de Bordeaux Service de néphrologie, Bordeaux
  - CHU Caen service de néphrologie, Caen
  - CHU Lyon service de néphrologie, Lyon
  - CHU Marseille Service de néphrologie, Marseille
  - CHU de Montpellier Hôpital Lapeyronie Service de Néphrologie, Montpellier
  - CHU de Nice Service de néphrologie, Nice
  - Hôpital Tenon Service de Nephrologie, Paris
  - Hôpital Européen Georges Pompidou Service de Nephrologie, Paris
  - CHU Reims service de néphrologie, Reims
  - CHU St Etienne Hopital Nord Service de néphrologie, Saint-Etienne
  - Clinique du Landy Centre de dialyse, Saint-Ouen
  - Néphrologie - Dialyse Centre de Rein Artificiel, Tassin-la-Demi-Lune
  - CH Valenciennes hémodialyse, Valenciennes
  - CHU de Nancy service de néphrologie, Vandeuvre Les Nancy

REFERENCES:
- [Background] Voormolen N, Noordzij M, Grootendorst DC, Beetz I, Sijpkens YW, van Manen JG, Boeschoten EW, Huisman RM, Krediet RT, Dekker FW; PREPARE study group. High plasma phosphate as a risk factor for decline in renal function and mortality in pre-dialysis patients. Nephrol Dial Transplant. 2007 Oct;22(10):2909-16. doi: 10.1093/ndt/gfm286. Epub 2007 May 21. PMID 17517792
- [Background] Levin A, Djurdjev O, Beaulieu M, Er L. Variability and risk factors for kidney disease progression and death following attainment of stage 4 CKD in a referred cohort. Am J Kidney Dis. 2008 Oct;52(4):661-71. doi: 10.1053/j.ajkd.2008.06.023. PMID 18805347
- [Background] Kestenbaum B, Sampson JN, Rudser KD, Patterson DJ, Seliger SL, Young B, Sherrard DJ, Andress DL. Serum phosphate levels and mortality risk among people with chronic kidney disease. J Am Soc Nephrol. 2005 Feb;16(2):520-8. doi: 10.1681/ASN.2004070602. Epub 2004 Dec 22. PMID 15615819
- [Background] Vassalotti JA, Uribarri J, Chen SC, Li S, Wang C, Collins AJ, Calvo MS, Whaley-Connell AT, McCullough PA, Norris KC; Kidney Early Evaluation Program Investigators. Trends in mineral metabolism: Kidney Early Evaluation Program (KEEP) and the National Health and Nutrition Examination Survey (NHANES) 1999-2004. Am J Kidney Dis. 2008 Apr;51(4 Suppl 2):S56-68. doi: 10.1053/j.ajkd.2007.12.018. PMID 18359409
- [Background] Danziger J. The bone-renal axis in early chronic kidney disease: an emerging paradigm. Nephrol Dial Transplant. 2008 Sep;23(9):2733-7. doi: 10.1093/ndt/gfn260. Epub 2008 May 9. No abstract available. PMID 18469306
- [Background] Inaba M, Okuno S, Imanishi Y, Yamada S, Shioi A, Yamakawa T, Ishimura E, Nishizawa Y. Role of fibroblast growth factor-23 in peripheral vascular calcification in non-diabetic and diabetic hemodialysis patients. Osteoporos Int. 2006 Oct;17(10):1506-13. doi: 10.1007/s00198-006-0154-6. Epub 2006 Aug 5. PMID 16896512
- [Background] Fliser D, Kollerits B, Neyer U, Ankerst DP, Lhotta K, Lingenhel A, Ritz E, Kronenberg F; MMKD Study Group; Kuen E, Konig P, Kraatz G, Mann JF, Muller GA, Kohler H, Riegler P. Fibroblast growth factor 23 (FGF23) predicts progression of chronic kidney disease: the Mild to Moderate Kidney Disease (MMKD) Study. J Am Soc Nephrol. 2007 Sep;18(9):2600-8. doi: 10.1681/ASN.2006080936. Epub 2007 Jul 26. PMID 17656479
- [Background] Gutierrez OM, Mannstadt M, Isakova T, Rauh-Hain JA, Tamez H, Shah A, Smith K, Lee H, Thadhani R, Juppner H, Wolf M. Fibroblast growth factor 23 and mortality among patients undergoing hemodialysis. N Engl J Med. 2008 Aug 7;359(6):584-92. doi: 10.1056/NEJMoa0706130. PMID 18687639
- [Background] Jean G, Terrat JC, Vanel T, Hurot JM, Lorriaux C, Mayor B, Chazot C. High levels of serum fibroblast growth factor (FGF)-23 are associated with increased mortality in long haemodialysis patients. Nephrol Dial Transplant. 2009 Sep;24(9):2792-6. doi: 10.1093/ndt/gfp191. Epub 2009 Apr 25. PMID 19395730
- [Background] Peiskerova M, Kalousova M, Kratochvilova M, Dusilova-Sulkova S, Uhrova J, Bandur S, Malbohan IM, Zima T, Tesar V. Fibroblast growth factor 23 and matrix-metalloproteinases in patients with chronic kidney disease: are they associated with cardiovascular disease? Kidney Blood Press Res. 2009;32(4):276-83. doi: 10.1159/000243050. Epub 2009 Oct 1. PMID 19797911
- [Background] JP Cristol, AS Bargnoux, AM Dupuy, M Morena, A Avignon and B Canaud. Biological markers of vascular calcifications in uremia. Médecine Nucléaire 2009; 33, 53-61.
- [Background] Stubbs JR, Quarles LD. Fibroblast growth factor 23: uremic toxin or innocent bystander in chronic kidney disease? Nephrol News Issues. 2009 May;23(6):33-4, 36-7. PMID 19534362
- [Background] Westerberg PA, Linde T, Wikstrom B, Ljunggren O, Stridsberg M, Larsson TE. Regulation of fibroblast growth factor-23 in chronic kidney disease. Nephrol Dial Transplant. 2007 Nov;22(11):3202-7. doi: 10.1093/ndt/gfm347. Epub 2007 Jun 13. PMID 17567652
- [Background] Shigematsu T, Kazama JJ, Yamashita T, Fukumoto S, Hosoya T, Gejyo F, Fukagawa M. Possible involvement of circulating fibroblast growth factor 23 in the development of secondary hyperparathyroidism associated with renal insufficiency. Am J Kidney Dis. 2004 Aug;44(2):250-6. doi: 10.1053/j.ajkd.2004.04.029. PMID 15264182
- [Background] Tanaka H, Hamano T, Fujii N, Tomida K, Matsui I, Mikami S, Nagasawa Y, Ito T, Moriyama T, Horio M, Imai E, Isaka Y, Rakugi H. The impact of diabetes mellitus on vitamin D metabolism in predialysis patients. Bone. 2009 Nov;45(5):949-55. doi: 10.1016/j.bone.2009.07.016. Epub 2009 Jul 23. PMID 19631779
- [Background] Urena Torres P, Friedlander G, de Vernejoul MC, Silve C, Prie D. Bone mass does not correlate with the serum fibroblast growth factor 23 in hemodialysis patients. Kidney Int. 2008 Jan;73(1):102-7. doi: 10.1038/sj.ki.5002622. Epub 2007 Oct 17. PMID 17943081
- [Background] Nagano N, Miyata S, Abe M, Kobayashi N, Wakita S, Yamashita T, Wada M. Effect of manipulating serum phosphorus with phosphate binder on circulating PTH and FGF23 in renal failure rats. Kidney Int. 2006 Feb;69(3):531-7. doi: 10.1038/sj.ki.5000020. PMID 16395276
- [Background] Oliveira RB, Cancela AL, Graciolli FG, Dos Reis LM, Draibe SA, Cuppari L, Carvalho AB, Jorgetti V, Canziani ME, Moyses RM. Early control of PTH and FGF23 in normophosphatemic CKD patients: a new target in CKD-MBD therapy? Clin J Am Soc Nephrol. 2010 Feb;5(2):286-91. doi: 10.2215/CJN.05420709. Epub 2009 Nov 12. PMID 19965540
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD-MBD Work Group. KDIGO clinical practice guideline for the diagnosis, evaluation, prevention, and treatment of Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD). Kidney Int Suppl. 2009 Aug;(113):S1-130. doi: 10.1038/ki.2009.188. PMID 19644521
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, Kusek JW, Van Lente F; Chronic Kidney Disease Epidemiology Collaboration. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med. 2006 Aug 15;145(4):247-54. doi: 10.7326/0003-4819-145-4-200608150-00004. PMID 16908915
- [Result] Liabeuf S, Ryckelynck JP, El Esper N, Urena P, Combe C, Dussol B, Fouque D, Vanhille P, Frimat L, Thervet E, Mentaverri R, Prie D, Choukroun G; FRENCH Study collaborators. Randomized Clinical Trial of Sevelamer Carbonate on Serum Klotho and Fibroblast Growth Factor 23 in CKD. Clin J Am Soc Nephrol. 2017 Dec 7;12(12):1930-1940. doi: 10.2215/CJN.03030317. Epub 2017 Oct 26. PMID 29074818
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086